CLINICAL TRIAL: NCT06167473
Title: Efficacy and Safety of Different Dosage of Umbilical Cord-mesenchymal Stem Cells Through Peripheral Vein in Patients With End-stage Liver Diseases
Brief Title: Effect of Different Dosage of Umbilical Cord-mesenchymal Stem Cells Through Peripheral Vein in Patients With ESLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHNKKY-DDSC
Record Dates: First submitted 2023-11-23; First posted 2023-12-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: End-stage Liver Diseases
Keywords: cirrhosis; end-stage liver diseases; umbilical cord-mesenchymal stem cells; randomized controlled trial
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Intervention Model Description: Before enrollment, all patients and/or their relatives will be informed about the study protocol, and sign the written informed consent forms. Eligible patients are randomly assigned at a ratio of 1:1 to low-dose stem cell group (1×10^6cells/kg per infusion) and a medium-high-dose stem cell group (3×10^6cells/kg per infusion).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low-dose stem cell group (1×10^6cells/kg per infusion) (Experimental): Peripheral intravenous infusion of low-dose stem cells
  Interventions: Biological: umbilical cord-mesenchymal stem cells
- medium-high-dose stem cell group (3×10^6cells/kg per infusion) (Experimental): Peripheral intravenous infusion of medium-high-dose stem cells
  Interventions: Biological: umbilical cord-mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord-mesenchymal stem cells — Different dosage of umbilical cord-mesenchymal stem cells through peripheral vein
  Other Names: UC-MSCs

SUMMARY:
There is a rise in the prevalence of end-stage liver disease during the last decade. End-stage liver disease has become one of the leading causes of death in Western countries. Liver transplantation is the only curative treatment for patients with end-stage liver disease. However, the shortage of donor, high cost, and postoperative complications limit its wide application in clinical practice. At present, stem cell-based therapy has been developed as an alternative treatment for end-stage liver disease. Stem cells can be differentiated into a variety of cell types, and stem cell transplantation, mainly umbilical cord-mesenchymal stem cells, has attracted more and more attention in the treatment of end-stage liver disease. The investigators therefore conduct a randomised controlled trial to investigate the efficacy and safety of human umbilical cord tissue mesenchymal stem cells for the treatment of end-stage liver disease.

DETAILED DESCRIPTION:
Twenty-two subjects with end-stage liver disease attending the Department of Gastroenterology of the General Hospital of the Northern Theatre of Operations are expected to be enrolled over a period of 1 year. The participants will be randomly divided into a low-dose stem cell group (1×10^6cells/kg per infusion) and a medium-high-dose stem cell group (3×10^6cells/kg per infusion), which are infused by peripheral vein. The investigators will observe ALT, AST, ALP, TBIL, ALB, PT, INR, MELD score, and Child-Pugh score in patients at weeks 1, 4, 8, 12, 24, and 48 post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. End-stage liver disease
3. Sign informed consent

Exclusion Criteria:

1. Tumours of the liver or other organs
2. Liver transplantation recipients
3. Acute myocardial infarction, acute heart failure, type I and type II respiratory failure, pulmonary embolism, acute cerebral infarction, acute cerebral haemorrhage and other serious cardiopulmonary diseases
4. Other diseases that may seriously affect the survival
5. Human immunodeficiency syndrome
6. Interferon or glucocorticoid therapy within 1 year
7. Treated for mental illness
8. Participation in other clinical trials within 30 days
9. Pregnant or breastfeeding subjects
10. Allergic asthma, allergic urticaria, eczema, or a history of multiple drug and food allergies
11. Other circumstances that are unsuitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 1 year
  Number of subjects surviving after one year

SECONDARY OUTCOMES:
Changes in liver function | 1, 4, 8, 12, 24, and 48 weeks
  The values of alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, serum albumin, prothrombin time, and international normalized ratio and the scores of MELD and Child-Pugh
Incidence of hepatic decompensation events | 1 year
  Number of patients who developed gastrointestinal bleeding, ascites and hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Mengfan Ruan, MM, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Ma XJ, Fei YY, Han HT, Xu J, Cheng L, Li X. Stem cell therapy in liver regeneration: Focus on mesenchymal stem cells and induced pluripotent stem cells. Pharmacol Ther. 2022 Apr;232:108004. doi: 10.1016/j.pharmthera.2021.108004. Epub 2021 Sep 28. PMID 34597754
- [Background] Khan S, Khan RS, Newsome PN. Cell Therapy for Liver Disease: From Promise to Reality. Semin Liver Dis. 2020 Nov;40(4):411-426. doi: 10.1055/s-0040-1717096. Epub 2020 Dec 24. PMID 33764490
- [Background] Alfaifi M, Eom YW, Newsome PN, Baik SK. Mesenchymal stromal cell therapy for liver diseases. J Hepatol. 2018 Jun;68(6):1272-1285. doi: 10.1016/j.jhep.2018.01.030. Epub 2018 Feb 7. PMID 29425678